CLINICAL TRIAL: NCT02244255
Title: An Eleven-Week, Open-Label, Randomized, Multicenter, Parallel-Design, Placebo Lead-in Study of FLOMAX® Capsules, 0.4 mg Daily Versus HYTRIN® Capsules, 5 mg (With Titration) Daily in Patients With the Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: FLOMAX® Versus HYTRIN® in Patients With the Signs and Symptoms of Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 527.17
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

ARMS (2):
- FLOMAX® (Experimental)
  Interventions: Drug: FLOMAX® capsules
- HYTRIN® (Active Comparator)
  Interventions: Drug: Ascending doses of HYTRIN® capsules

INTERVENTIONS:
Drug: FLOMAX® capsules
  Other Names: Tamsulosin hydrochloride
  Arms: FLOMAX®
Drug: Ascending doses of HYTRIN® capsules
  Arms: HYTRIN®

SUMMARY:
1. To study the early onset of symptomatic relief afforded by FLOMAX® capsules, 0.4 mg daily as compared to HYTRIN® capsules, 5 mg (with titration) daily in patients with the signs and symptoms of benign prostatic hyperplasia (BPH)
2. To evaluate patient's tolerability to the use of FLOMAX® capsules 0.4 mg daily in comparison to HYTRIN® capsules, 5 mg (with titration) daily for the treatment of the symptoms of benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Male patients (45 years of age or older) diagnosed with benign prostatic hyperplasia
* Patients with a total score on the AUA Symptom Index for BPH of at least 13 points at each of the three initial visits (Visits 1, 2 and 3)
* A baseline prostate specific antigen (PSA) of ≤ 4.0 ng/ml
* Patients who are able to give written informed consent before performing screening examinations or tests
* Patients being judged by the investigator to be reliable and able to follow protocol procedures (including the return visits schedule), and cooperate in the completion of tests related to safety and efficacy

Exclusion Criteria:

* Patients with a history of an allergy to alpha blockers, alpha/beta blockers or patients who have had a "first dose hypotensive episode" upon starting therapy with an alpha blocker
* Patients who are currently being treated or who, in the last 3 months, have been treated with finasteride
* Participated in an investigational drug study within 4 weeks prior to starting placebo phase
* Patients taking medication in the following classes and unable to discontinue them at least two weeks before the study and for the duration of the study

  * Alpha adrenergic blocking agents
  * Alpha adrenergic agonists
  * Drugs with anticholinergic activity (including antihistamines)
  * Antispasmodics
  * Parasympathomimetics and cholinomimetics
* Peripheral or central neurologic disease including, but not limited to, transient ischemic attacks, stroke, dementia, multiple sclerosis, spinal cord injury, recurrent episodes of dizziness, vertigo, or loss of consciousness, clinically evident diabetic neuropathy, brain and/or spinal cord tumors
* History of a pathological fall (unintentional change in body position) occurring under circumstances in which normal homeostatic mechanisms would ordinarily maintain stability, or syncope during the last year
* More than one episode of angina within the past 6 months
* Ambulation requiring assistance (i.e., canes, walkers, etc.)
* Documented myocardial infarction (by ECG) within the past 6 months or evidence of a myocardial infarction on ECG whose age cannot be determined
* New York Heart Association Class III or IV congestive heart failure
* Prosthetic heart valves, cardiac devices or prior history of endocarditis
* Clinically significant cardiac arrhythmias either diagnosed by ECG or recorded in the medical history, whether or not accompanied by symptoms (e.g., dizziness, presyncope, syncope, unsteadiness)
* Infravesical obstruction by history due to:

  * Vesical neck contracture
  * Clinical suspicion of prostate carcinoma
  * Mullerian duct cysts
  * Urethral obstruction due to stricture, valves, sclerosis or urethral tumor
  * Inflammatory or infectious conditions
  * Detrusor-sphincter dyssynergia
* Prior transurethral resection of the prostate (TURP) or open prostatectomy
* History of instrumentation of the urinary tract (cytoscopy or catheterization) within 30 days prior to the start of the study
* Prior pelvic surgery for malignancy or bowel resection
* History or diagnosis of genitourinary malignancy
* History of an episode of acute urinary retention within three months prior to the start of the study. (Urinary retention is to be considered acute if the patient has to be sent to a hospital for catheterization)
* Patients with the current diagnosis of either bladder, ureter, or kidney stones
* Patients with a current diagnosis of suspected prostatitis
* Patients with a history of a neurogenic bladder
* Urinary tract infection (i.e., positive urine culture) yielding pathogenic bacteria > 10**5 colony forming units (CFU) per milliliter in a properly obtained clean voided urine specimen which has been properly cultured or a laboratory report of a urinary tract infection or signs/symptoms indicative of a urinary tract infection such as [increased WBC's in the urine (15-30 white blood cells (WBC)/high powered field), dysuria, costovertebral tenderness, and urinary frequency accompanied by fever] within four weeks of baseline (Visit 3)
* Evidence of significant renal dysfunction based upon a serum creatinine greater than two times the upper limit of normal levels established by the central laboratory used in this study
* Laboratory tests during the screening phase:

  * Hemoglobin: < 12.0 g/dL
  * Leukocytes: < 3000/mm3
  * Liver Enzymes: (serum glutamic oxaloacetic transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT), and alkaline phosphatase): more than two times the upper limit of normal levels established by the central laboratory used in the study
* Clinically relevant conditions which might interfere with the patient's ability to participate in the study including, but not limited to, the following: neurologic, gastrointestinal, cardiovascular including uncontrolled hypertension defined as a sitting diastolic blood pressure ≥ 95 mmHg with or without treatment, hepatic, renal, psychiatric, hematologic or respiratory disease, clinically relevant laboratory abnormalities based upon the investigator's judgment
* Hypertensive patients initially using HYTRIN® as a monotherapy for both hypertension and BPH
* Patients with cancer or diagnosis of cancer within five years of baseline
* Patients who have been receiving cimetidine, warfarin, or herbal medications specifically for treatment of any urological problems within four weeks prior to the baseline
* Patients who show poor compliance in the initial placebo period by:

  * not returning unused medication bottles for Visits 2 or 3
  * having taken < 80% or > 120% of prescribed doses during any visit interval between Visit (1, 2 or 3)
* Postural symptoms during the initial placebo period, e.g., lightheadedness (on more than three occasions), fainting, blurring or loss of vision, profound weakness, or unsteadiness, with or without a change in blood pressure and/or pulse rate
* Patients with poorly controlled diabetes mellitus (urine positive for glucose (> 1+) on each of 2 urinalyses during the placebo evaluation period)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1993 (Actual)
Dates: Start 1998-08; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Changes in American Urological Association (AUA) symptom score index | Pre-dose, up to day 57 after start of treatment

SECONDARY OUTCOMES:
Changes in AUA bother score index | Pre-dose, up to 57days after start of treatment
  Validated quality of life questionnaire for urinary problems containing:
  * AUA obstructive symptom score
  * AUA irritative symptom score
  * AUA nocturia symptom score
Changes in BPH impact index score | Pre-dose, up to 57 days after start of treatment
Global assessment by investigator on a 5-point scale | Day 5, up to day 57 after start of treatment
Number of patients with clinically relevant changes from baselinein laboratory values | Pre-dose, day 57 after start of treatment
Number of patients with clinically significant changes in vital signs | Pre-dose, up to 57 days after start of treatment
Number of patients with clinically relevant changes from baseline in ECG | Pre-dose, up to 57 days after start of treatment
Number of patients with adverse events | Up to day 57